CLINICAL TRIAL: NCT06042257
Title: Guanfacine for Hyperactivity in Children With Down Syndrome (HYPEbeGONE_DS)
Acronym: HYP01
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was stopped after careful review of product manufacturing needs and available resources. Decision reflects consideration of feasibility, enrollment challenges, and overall program goals.
Sponsor: Rachel G. Greenberg, MD, MB, MHS (Other)
Collaborators: The Emmes Company, LLC (Industry); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor-Investigator, Rachel G. Greenberg, MD, MB, MHS, Associate Professor of Pediatrics, Duke University
Organization: Duke University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Pro00111256; HHSN275201800003I (Other Grant/Funding Number: National Institute of Child Health and Human Development)
Record Dates: First submitted 2023-07-31; First posted 2023-09-18 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-01

CONDITIONS: Hyperactivity in Children With Down Syndrome; Impulsivity in Children With Down Syndrome
Keywords: hyperactivity; impulsivity; inattention
MeSH Terms: conditions — Spasm; Impulsive Behavior | interventions — Guanfacine

STUDY DESIGN:
Intervention Model Description: Participants will be randomized 2:1 to GIR or placebo.
Who Masked: Participant, Care Provider, Investigator
Masking Description: A masked investigational pharmacist or designee will dispense study product according to randomization treatment assignments. All other site staff as well as participants and parents/legal guardians will also be masked for up to 8 weeks while the study participant is receiving study product.
  Participants, parents/legal guardians, site staff, and study administrators will be unmasked at the 8 week study visit.
  Emergency unmasking may occur at any time throughout the study in the event that knowledge of the actual treatment is absolutely essential for further management of the participant.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Guanfacine Hydrochloride Immediate Release (Active Comparator): Eligible participants will receive GIR for up to 8 weeks. The treatment period will consist of study product administration from day 0 through day 56 with a masked dose-escalation period from day 0 through day 49.
  Interventions: Drug: Guanfacine Hydrochloride Immediate Release
- Placebo (Placebo Comparator): Eligible participants will receive Placebo for up to 8 weeks.The treatment period will consist of study product administration from day 0 through day 56 with a masked dose-escalation period from day 0 through day 49.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Guanfacine Hydrochloride Immediate Release — 0.5 mg capsules
  Arms: Guanfacine Hydrochloride Immediate Release
Drug: Placebo — Matching placebo capsule
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine efficacy of guanfacine immediate release (GIR) for the treatment of hyperactivity/impulsivity and inattention in children 6-12 years of age with Down syndrome (DS) after 8 weeks of treatment.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled flexibly dosed trial of guanfacine immediate release (GIR) in children with Down syndrome (DS) and symptoms of hyperactivity, inattention, and impulsivity. Participants will undergo a screening period of up to 29 days. Eligible participants meeting study criteria will be randomized 2:1 GIR or placebo. There are a total of up to 4 in person visits (screening, baseline, at Week 4, and at Week 8). Participants will receive GIR or placebo for up to 8 weeks. Weekly dose escalation will be determined via a telephone assessment at Weeks 1-3 and Weeks 4-7. Unmasking of participant and site staff will occur at the week 8, in-person visit. After unmasking, participants who were randomized to receive GIR will be given the option to 1) remain on GIR and to transition to open-label GIR per standard of care or 2) taper off of GIR. A Telephone Safety Assessment will be conducted for all participants, at 5 (+2) days after final study product administration. Blood specimens will be collected at the Week 4 and Week 8 visits for Pharmacokinetic (PK) analyses and lab assessments. Participants will be asked to keep a daily study diary and will complete study measures at screening/baseline, Week 4 and Week 8. Parents/Caregivers will need to complete the Study Diary during the bridge/taper period for those who are in the GIR arm.

ELIGIBILITY:
Inclusion:

1. Parent/Legal Guardian can understand the consent process and is willing to provide informed consent/HIPAA authorization prior to the conduct of any study-related procedures. When applicable, the minor participant is willing to provide assent.
2. Participant has clinical diagnosis of non-mosaic DS.
3. Participant is between 6 and 12 years of age (inclusive) at time of consent.
4. Participant weight is ≥ 25 kg.
5. Participant has clinically significant symptoms of hyperactivity, inattention and impulsivity manifested as minimum scores of the following rating scales within 30 days of randomization:

   1. A minimum score of 18 on the parent-reported ABC-H subscale, AND
   2. A minimum score of moderate or greater (≥ 4) on the clinician reported Clinical Global Impression Severity (CGI-S) score specific to hyperactivity, inattention and impulsivity behaviors.
6. Participant has co-morbid medical screening and clearance to proceed with a non-stimulant medication trial with GIR within 30 days of randomization.
7. Participant is willing and able to comply with study procedures, including adherence to medication dosing schedule.

Exclusion:

1. Participant has received guanfacine (any formulation) within 30 days of randomization.
2. Participant has received any of the following concomitant medication classes within 30 days of randomization:

   1. Strong CYP3A4 inhibitors (e.g., boceprevir, clarithromycin, conivaptan, grapefruit juice, indinavir, itraconazole, ketoconazole, lopinavir/ritonavir, mibefradil, nefazodone, nelfinavir, posaconazole, ritonavir, saquinavir, telaprevir, telithromycin, and voriconazole)
   2. Strong CYP3A4 inducers (e.g., avasimibe, carbamazepine, phenytoin, rifampin, and St. John's wort)
3. Participant has a psychiatric comorbidity, such as major depressive disorder, bipolar disorder, obsessive-compulsive disorder, or a psychotic disorder, that requires a pharmacological treatment other than guanfacine
4. For participants ≥ 8 years old at the time of consent, participant has a history of suicidality or positive screen on Ask Suicide-Screening Questions (asQ) Tool.
5. Participant is currently in or plans to participate in another interventional study.
6. Participant has a known hypersensitivity to guanfacine.
7. Participant has had a previous guanfacine treatment failure, as determined by their primary treating physician.
8. Participant has had a change in another medication intended to treat symptoms of hyperactivity, inattention, and impulsivity within the last 2 weeks.
9. Participant has had a seizure within the last 6 months.
10. Participant has had a change in their anti-convulsant dose within the last 4 weeks.
11. Participant has a cardiac-related condition including:

    1. Significant symptomatic bradycardia;
    2. 2nd degree or 3rd degree (complete) heart block;
    3. Baseline heart rate (HR) or systolic blood pressure (BP) > 2 standard deviations (SD) below mean for age as determined by medical examination;
    4. History of aborted sudden cardiac death, unexplained syncope or near syncope, or historical use of a pacemaker as determined by medical history will require clearance by cardiology prior to enrollment;
    5. Known history of congenital heart disease which requires ongoing care for monitoring or management will require clearance by cardiology prior to enrollment.
12. Participant has a history of untreated severe obstructive sleep apnea defined as obstructive apnea hypopnea index (OAHI) ≥ 10 events per hour or aortic regurgitation (AR). Participants with an OAHI index > 10/hr are eligible if managed with continuous positive airway pressure (CPAP).
13. Participant has untreated thyroid disease.
14. Participant has a known hepatic impairment defined as aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 2x the upper limit of normal (ULN) for age.
15. Participant has known impending or renal failure defined as:

    1. Anuria diagnosed within 12 hours prior to enrollment;
    2. Requiring renal replacement therapy.
16. Participant is pregnant.
17. Participant has any condition which would make the participant, in the opinion of the investigator, unsuitable for the study.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 3 (Actual)
Dates: Start 2024-12-09 (Actual); Primary Completion 2025-05-17 (Actual); Study Completion 2025-08-12 (Actual)

PRIMARY OUTCOMES:
Change in parent-rated ABC-H (Aberrant Behavior Checklist-Hyperactivity) subscale core | Baseline to Week 8
  Change from baseline to Week 8 of the ABC-H subscale score. The ABC-H is a subscale of the ABC. Each of the 16 items is scored as 0 (never a problem), 1 (slight problem), 2 (moderately serious problem), or 3 (severe problem). The total score range is 0 to 48, where a higher score indicates endorsement of greater hyperactivity. Rating based on patient's behavior in last 4 weeks.

SECONDARY OUTCOMES:
Change in parent-rated ABC-H (Aberrant Behavior Checklist-Hyperactivity) subscale core | Baseline to Week 4
  Change from baseline to Week 4 of the ABC-H subscale score. The ABC-H is a subscale of the ABC. Each of the 16 items is scored as 0 (never a problem), 1 (slight problem), 2 (moderately serious problem), or 3 (severe problem). The total score range is 0 to 48, where a higher score indicates endorsement of greater hyperactivity. Rating based on patient's behavior in last 4 weeks.
Proportion of participants with a CGI-I (Clinical Global Impression-Improvement) score of 2 or better at Week 4 | Baseline to Week 4
  CGI-I specific to hyperactivity, inattention and impulsivity behaviors. The CGI-I is a seven-point scale that requires the clinician to assess how much the patient's illness has improved or worsened relative to a baseline state at the beginning of the intervention. 1 = Very much improved, 2 = Much improved, 3 = Minimally improved, 4 = No change, 5 = Minimally worse, 6 = Much worse, 7 = Very much worse.
Proportion of participants with a CGI-I (Clinical Global Impression-Improvement) score of 2 or better at Week 8 | Baseline to Week 8
  CGI-I specific to hyperactivity, inattention and impulsivity behaviors. The CGI-I is a seven-point scale that requires the clinician to assess how much the patient's illness has improved or worsened relative to a baseline state at the beginning of the intervention. 1 = Very much improved, 2 = Much improved, 3 = Minimally improved, 4 = No change, 5 = Minimally worse, 6 = Much worse, 7 = Very much worse.
Safety of GIR (guanfacine immediate release) | Baseline through Week 8
  Number of participants with adverse events (AEs), serious adverse events (SAEs), or events of special interest (ESIs).

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Greenberg, Principal Investigator — DCRI
Locations (15):
- United States (15):
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - Yale University School of Medicine, New Haven, Connecticut
  - Emory University, Atlanta, Georgia
  - Ann and Robert H. Lurie Hospital of Chicago, Chicago, Illinois
  - University of Iowa, Iowa City, Iowa
  - Kennedy Krieger Institute, Baltimore, Maryland
  - Boston Children's Hospital, Boston, Massachusetts
  - Massachusetts General Hospital, Lexington, Massachusetts
  - Atrium Health-Wake Forest School of Medicine, Charlotte, North Carolina
  - Duke University Hospital, Durham, North Carolina
  - Akron Children's Hospital, Akron, Ohio
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - Virginia Center for Children, Richmond, Virginia
  - University of Washington, Seattle, Washington
  - University of Wisconsin Madison, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
All data collected is uploaded into the National Institute of Health Data Repository (DASH) at the end of the study (de-identified).
Supporting Information: Study Protocol, ICF
Time Frame: Data will be uploaded to the repository within 2 years of study completion. It will be maintained in the repository indefinitely.
Access Criteria: In order to have access, researchers have to complete a Data access request. NICHD will review the request and either approve or deny it. IRB approval must be obtained by the researcher to access the data.
  https://dash.nichd.nih.gov/Resource/DataRequestChecklist
URL: https://dash.nichd.nih.gov

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-08-29): https://cdn.clinicaltrials.gov/large-docs/57/NCT06042257/Prot_SAP_000.pdf
  • Informed Consent Form (2023-11-06): https://cdn.clinicaltrials.gov/large-docs/57/NCT06042257/ICF_001.pdf